CLINICAL TRIAL: NCT07033442
Title: Effects Of Inhalation Anaesthesia and Total Intravenous Anaesthesia on Intraocular Pressure in Robotic Prostate Surgery
Brief Title: Effects Of Anaesthesia on Intraocular Pressure in Robotic Prostate Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Aysun Erşen Yüngül, Principal Investigator, Ataturk Training and Research Hospital
Allocation: Randomized | Model: Parallel | Purpose: Other
Other Study IDs: EthicsApproval: 152
Record Dates: First submitted 2025-05-19; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Anaesthesia; Intraocular Pressure; Trendelenburg Position; Robot Assisted Laparoscopic Radical Prostatectomy; Total Intravenous Anesthesia; Inhalation Anesthesia
Keywords: Robot Assisted Laparoscopic Radical prostatectomy; Intraoculer Pressure; Total Intravenous Anesthesia; Inhalation Anaesthesia
MeSH Terms: interventions — Sevoflurane; Propofol; Remifentanil; Rocuronium; Thiopental; Injections; Atropine; Intraocular Pressure; Respiration, Artificial; Crystalloid Solutions; Intubation, Intratracheal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- This group received general anesthesia maintained with an inhalation-based technique. (Active Comparator): Anesthesia was maintained in the patients using sevoflurane+remifentail infusion in Arm 1
  Interventions: Drug: Sevoflurane (Volatile Anesthetic); Drug: Remifentanil 2 MG; Drug: Rocuronium 50 mg/5 ml; Drug: Lidocaine %2 ampoule; Drug: Thiopental 500 mg vial for injection; Drug: Neostigmine 0,5 mg/ml ampoule; Drug: Atropine Sulphate 0.5mg/ml ampoule; Drug: Ephedrine Hydrochloride 0,05 mg/ml ampoule; Procedure: CO₂ Pneumoperitoneum; Device: Bispectral index (BIS) Monitoring; Procedure: intraocular pressure measurement; Procedure: intraarterial cannulation and pressure measurement; Procedure: Mechanical Ventilation; Procedure: Peripheral Intravenous Cannulation; Drug: Crystalloid solutions; Procedure: Endotracheal Intubation; Procedure: American Society of Anesthesiologists (ASA) Standard Monitors; Procedure: Ventilatory Pressure and Compliance Monitoring
- This group received general anesthesia maintained with a total intravenous technique. (Active Comparator): Anesthesia was maintained in the patients using propofol+remifentanil infusion in Arm 2
  Interventions: Drug: Propofol 1%; Drug: Remifentanil 2 MG; Drug: Rocuronium 50 mg/5 ml; Drug: Lidocaine %2 ampoule; Drug: Neostigmine 0,5 mg/ml ampoule; Drug: Atropine Sulphate 0.5mg/ml ampoule; Drug: Ephedrine Hydrochloride 0,05 mg/ml ampoule; Procedure: CO₂ Pneumoperitoneum; Device: Bispectral index (BIS) Monitoring; Procedure: intraocular pressure measurement; Procedure: intraarterial cannulation and pressure measurement; Procedure: Mechanical Ventilation; Procedure: Peripheral Intravenous Cannulation; Drug: Crystalloid solutions; Procedure: Endotracheal Intubation; Procedure: American Society of Anesthesiologists (ASA) Standard Monitors; Procedure: Ventilatory Pressure and Compliance Monitoring

INTERVENTIONS:
Drug: Sevoflurane (Volatile Anesthetic) — Inhalational anesthetic used for maintenance of anesthesia. Administered at 2-3% concentration in a 40% oxygen-air mixture to maintain BIS values between 40-60.
  Arms: This group received general anesthesia maintained with an inhalation-based technique.
Drug: Propofol 1% — Intravenous hypnotic agent used for induction (2-3 mg/kg) and maintenance (50-150 μg/kg/min) of anesthesia. Titrated to maintain BIS values between 40-60.
  Arms: This group received general anesthesia maintained with a total intravenous technique.
Drug: Remifentanil 2 MG — Short-acting opioid used for induction and maintenance of anesthesia at a dose of 1 μg/kg IV (induction) and 0.05-0.25 μg/kg/min (maintenance).
Drug: Rocuronium 50 mg/5 ml — Neuromuscular blocker administered IV at 0.6-1.2 mg/kg for induction and 0.15 mg/kg for maintenance of muscle relaxation during surgery.
Drug: Lidocaine %2 ampoule — Administered intravenously at 1-1.5 mg/kg before anesthesia induction to reduce injection pain and facilitate induction.
Drug: Thiopental 500 mg vial for injection — Intravenous anesthetic agent used for induction of anesthesia at 4-6 mg/kg.
  Arms: This group received general anesthesia maintained with an inhalation-based technique.
Drug: Neostigmine 0,5 mg/ml ampoule — Administered IV at 0.04 mg/kg for reversal of neuromuscular blockade at the end of the procedure.
Drug: Atropine Sulphate 0.5mg/ml ampoule — Administered intravenously (0.4 mg per 1 mg neostigmine) to counteract muscarinic effects during neuromuscular blockade reversal; also 0.5 mg IV in cases of intraoperative bradycardia (HR < 45 bpm).
Drug: Ephedrine Hydrochloride 0,05 mg/ml ampoule — Used intravenously at 0.1 mg/kg to manage intraoperative hypotension unresponsive to fluid and anesthetic dose adjustment.
Procedure: CO₂ Pneumoperitoneum — Creation of pneumoperitoneum with CO₂ insufflation for robotic prostatectomy; monitoring and recording of intra-abdominal pressures.
Device: Bispectral index (BIS) Monitoring — Monitoring of depth of anesthesia using bispectral index values; frontal placement preoperatively and throughout surgery. BIS maintained between 40-60.
Procedure: intraocular pressure measurement — Measurement of intraocular pressure (IOP) in both eyes at multiple intraoperative and postoperative time points (T0-T9).
Procedure: intraarterial cannulation and pressure measurement — Invasive arterial blood pressure measurement and blood gas measurements via an 18G catheter inserted into the radial artery
Procedure: Mechanical Ventilation — Ventilation initiated after intubation with volume-controlled settings (TV 6-8 ml/kg, RR 12, FiO₂ 50%), adjusted to maintain ETCO₂ between 30-36 mmHg.
Procedure: Peripheral Intravenous Cannulation — All participants received peripheral intravenous cannulation using 18-20 G IV cannulas placed on the dorsum of the hand before anesthesia induction.
Drug: Crystalloid solutions — Participants received calculated maintenance fluids with crystalloids through intravenous infusion prior to and during surgery.
Procedure: Endotracheal Intubation — After induction of anesthesia and neuromuscular blockade, endotracheal intubation was performed using standard technique in all participants.
Procedure: American Society of Anesthesiologists (ASA) Standard Monitors — Routine ASA monitoring, including noninvasive blood pressure, ECG (D2 derivation), End-tidal carbon dioxide (ETCO₂) and Peripheral Oxygen Saturation (SpO₂), was performed in all patients, starting from the preoperative period and continuing throughout the surgery.
Procedure: Ventilatory Pressure and Compliance Monitoring — Throughout the procedure, the following lung mechanics were continuously measured: PEEP, peak airway pressure (PEAK), mean airway pressure (Pmean), plateau pressure (Pplato), and dynamic compliance.

SUMMARY:
Robot-assisted surgery is now commonly used to treat prostate cancer. This type of surgery, called robot-assisted prostatectomy, helps doctors operate more precisely and allows patients to heal faster. But there are some special things to be careful about during these surgeries.

During the operation, the patient is placed in a steep head-down position for a long time. Staying in this position for a long period can cause the pressure inside the eyes-called intraocular pressure (IOP)-to go up. High eye pressure can be risky, especially for people who already have eye problems.

This study looked at different types of anesthesia used during robotic prostate surgery to see how they affect eye pressure. The goal was to find out which type of anesthesia causes less of an increase in eye pressure.

DETAILED DESCRIPTION:
In this study, the aim was to investigate the effects of hemodynamic changes induced by the steep Trendelenburg position and pneumoperitoneum, surgical duration, blood gas parameters, and the type of anesthesia administered on intraocular pressure (IOP) during robotic prostatectomy.

Prostate cancer is the most common type of cancer among men. Among the various treatment options, robot-assisted radical prostatectomy (RARP) stands out as the most recent and technologically advanced surgical approach.

This randomized and prospective study was conducted at the operating rooms of Ankara Atatürk Training and Research Hospital following approval by the Ethics Committee. Sixty cooperative adult male patients scheduled to undergo robotic prostatectomy under general anesthesia and classified as ASA physical status I-II were enrolled in the study after providing informed written consent.

Patients with severe cardiac disease, restrictive or obstructive pulmonary disease, renal or hepatic insufficiency, a history of hypersensitivity to anesthetic agents, psychiatric disorders, neurologic diseases, previous intracranial surgery, chronic alcohol, sedative, tranquilizer, or analgesic use, glaucoma, or those receiving medications known to affect IOP, as well as patients predicted to present with difficult intubation on direct laryngoscopy, were excluded from the study.

Participants were randomly assigned to one of two groups by drawing a label from a sealed envelope: Group 1 received inhalation anesthesia, and Group 2 received total intravenous anesthesia (TIVA). Demographic data were recorded. Prior to the induction of general anesthesia, while the participants were in the supine position, baseline measurements were taken, including heart rate (HR), mean arterial pressure (MAP), peripheral oxygen saturation (SpO₂), end-tidal CO₂ (ETCO₂), bispectral index (BIS), and IOP in both eyes.

Anesthesia induction was carried out using the following agents: patients in Group 1 received intravenous Lidocaine at a dose of 1-1.5 mg/kg, Thiopental 4-6 mg/kg, Remifentanil 1 µg/kg, and Rocuronium 0.6-1.2 mg/kg. In Group 2, Lidocaine 1-1.5 mg/kg, Propofol 2-3 mg/kg, Remifentanil 1 µg/kg, and Rocuronium 0.6-1.2 mg/kg were administered. For anesthesia maintenance, Group 1 was managed with Sevoflurane combined with a Remifentanil infusion, while Group 2 received a combination of Propofol and Remifentanil infusions.

Intraocular pressure (IOP), hemodynamic parameters, arterial blood gas values, pulmonary mechanics, heart rate (HR), mean arterial pressure (MAP), systolic and diastolic blood pressure, bispectral index (BIS), peripheral oxygen saturation (SpO₂), and end-tidal carbon dioxide (ETCO₂) levels were evaluated at ten specific time points throughout the procedure. These included: before anesthesia induction (T0); 10 minutes after induction (T1); 2 minutes after positioning the participant in the steep Trendelenburg position (T2); 2 minutes following carbon dioxide (CO₂) insufflation (T3); 1 hour (T4), 2 hours (T5), and 3 hours (T6) after CO₂ insufflation; 2 minutes after CO₂ desufflation (T7); 2 minutes after returning the participant to the supine position (T8); and 45 minutes postoperatively (T9).

Intra-abdominal pressures generated by CO₂ insufflation, as well as the minimum alveolar concentration (MAC) of sevoflurane and ETCO₂ values, were also recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo robot-assisted prostate surgery with ASA I-II

Exclusion Criteria:

* serious cardiac disease
* restrictive and obstructive lung disease
* renal and hepatic insufficiency
* with a history of hypersensitivity to the agents to be used
* with psychiatric disorders
* with a history of neurological disease
* who had intracranial surgery
* with a history of alcohol, sedative, tranquilizer and long-term analgesic use,
* with glaucoma and those taking medications that would affect IOP
* who were thought to have difficult intubation during direct laryngoscopy.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-07-23 (Actual); Primary Completion 2015-11-17 (Actual); Study Completion 2015-12-24 (Actual)

PRIMARY OUTCOMES:
Intraocular Pressure Measured Using Tono-Pen at Multiple Perioperative Time Points (mmHg) | From 10 minutes before anesthesia induction to 45 minutes postoperatively
  Intraocular pressure (IOP) will be measured in both eyes using a handheld Tono-Pen tonometer at the following predefined perioperative time points:
  T0 (before anesthesia induction) T1 (10 minutes after induction) T2 (2 minutes after steep Trendelenburg positioning) T3 (2 minutes after carbon dioxide (CO₂) insufflation) T4 (1 hour after CO₂ insufflation) T5 (2 hours after CO₂ insufflation) T6 (3 hours after CO₂ insufflation) T7 (2 minutes after CO₂ desufflation) T8 (2 minutes after return to supine position) T9 (45 minutes postoperatively)
  The unit of measurement is mmHg at each time point. Each time point will be reported separately. To ensure consistency, all measurements will be performed by the same ophthalmologist.

SECONDARY OUTCOMES:
Heart Rate at Defined Perioperative Time Points (bpm) | From 10 minutes before anesthesia induction to 45 minutes postoperatively.
  Heart rate (HR) will be measured non-invasively using standard ASA monitoring equipment at the following perioperative time points:
  T0 (before anesthesia induction) T1 (10 minutes after induction) T2 (2 minutes after Trendelenburg positioning) T3 (2 minutes after carbon dioxide (CO₂) insufflation) T4 (1 hour after CO₂ insufflation) T5 (2 hours after CO₂ insufflation) T6 (3 hours after CO₂ insufflation) T7 (2 minutes after CO₂ desufflation) T8 (2 minutes after return to supine position) T9 (45 minutes postoperatively)
  Heart rate will be reported separately for each time point.
Bispectral Index Score (BIS) Values at Defined Perioperative Time Points | From 10 minutes before anesthesia induction to 45 minutes postoperatively.
  The Bispectral Index Score (BIS) will be monitored to assess the depth of anesthesia. The BIS scale ranges from 0 (deep coma) to 100 (fully awake). Lower scores indicate deeper anesthesia, while higher scores indicate lighter anesthesia or awareness. Bispectral Index Score (BIS) values will be continuously monitored using the BIS VISTA Monitor (Covidien REF 185-0151). BIS values will be recorded at the following predefined perioperative time points to assess anesthetic depth:
  T0 (before anesthesia induction) T1 (10 minutes after induction) T2 (2 minutes after Trendelenburg positioning) T3 (2 minutes after carbon dioxide (CO₂) insufflation) T4 (1 hour after CO₂ insufflation) T5 (2 hours after CO₂ insufflation) T6 (3 hours after CO₂ insufflation) T7 (2 minutes after CO₂ desufflation) T8 (2 minutes after return to supine position) T9 (45 minutes postoperatively) Each BIS value will be reported separately for each time point.
Intraabdominal Pressure (IAP) at Defined Perioperative Time Points (mmHg) | From CO₂ insufflation to desufflation during the intraoperative period.
  Intraabdominal pressure (IAP) will be monitored via the robotic insufflation system and recorded at the following predefined perioperative time points during carbon dioxide (CO₂) insufflation:
  T3 (2 minutes after CO₂ insufflation) T4 (1 hour after CO₂ insufflation) T5 (2 hours after CO₂ insufflation) T6 (3 hours after CO₂ insufflation) T7 (2 minutes after CO₂ desufflation)
  Each IAP measurement will be reported separately for each time point.
Peripheral Oxygen Saturation (SpO₂) at Defined Perioperative Time Points (%) | From 10 minutes before anesthesia induction to 45 minutes postoperatively.
  Description:
  Peripheral oxygen saturation (SpO₂) will be continuously monitored using pulse oximetry as part of standard ASA monitoring.
  SpO₂ values will be documented at the following predefined perioperative time points to assess oxygenation:
  T0 (before anesthesia induction) T1 (10 minutes after induction) T2 (2 minutes after Trendelenburg positioning) T3 (2 minutes after carbon dioxide (CO₂) insufflation) T4 (1 hour after CO₂ insufflation) T5 (2 hours after CO₂ insufflation) T6 (3 hours after CO₂ insufflation) T7 (2 minutes after CO₂ desufflation) T8 (2 minutes after returning to supine position) T9 (45 minutes postoperatively)
  Each SpO₂ measurement will be reported separately for each time point.
End-Tidal Carbon Dioxide (ETCO₂) Levels at Defined Perioperative Time Points (mmHg) | From 10 minutes before anesthesia induction to 45 minutes postoperatively.
  End-tidal carbon dioxide (ETCO₂) will be continuously measured through the ventilator (Mindray WATO EX-65) and documented at the following predefined perioperative time points:
  T0 (before anesthesia induction) T1 (10 minutes after induction) T2 (2 minutes after Trendelenburg positioning) T3 (2 minutes after carbon dioxide (CO₂) insufflation) T4 (1 hour after CO₂ insufflation) T5 (2 hours after CO₂ insufflation) T6 (3 hours after CO₂ insufflation) T7 (2 minutes after CO₂ desufflation) T8 (2 minutes after return to supine position) T9 (45 minutes postoperatively)
  Each ETCO₂ measurement will be reported separately for each time point.
Mean Arterial Pressure at Defined Perioperative Time Points (mmHg) | From 10 minutes before anesthesia induction to 45 minutes postoperatively.
  Mean arterial pressure (MAP) will be measured non-invasively using standard ASA monitoring equipment at the following perioperative time points:
  T0 (before anesthesia induction) T1 (10 minutes after induction) T2 (2 minutes after Trendelenburg positioning) T3 (2 minutes after carbon dioxide (CO₂) insufflation) T4 (1 hour after CO₂ insufflation) T5 (2 hours after CO₂ insufflation) T6 (3 hours after CO₂ insufflation) T7 (2 minutes after CO₂ desufflation) T8 (2 minutes after return to supine position) T9 (45 minutes postoperatively)
  Mean arterial pressure will be reported separately for each time point.
Arterial Partial Pressure of Oxygen (PaO₂) at Selected Perioperative Time Points (mmHg) | From 10 minutes before anesthesia induction to 45 minutes postoperatively.
  Arterial blood gas samples will be collected at the following perioperative time points to measure partial pressure of oxygen (PaO₂):
  T0 (before anesthesia induction) T1 (10 minutes after induction) T2 (2 minutes after Trendelenburg positioning) T3 (2 minutes after carbon dioxide (CO₂) insufflation) T4 (1 hour after CO₂ insufflation) T5 (2 hours after CO₂ insufflation) T6 (3 hours after CO₂ insufflation) T7 (2 minutes after CO₂ desufflation) T8 (2 minutes after return to supine position) T9 (45 minutes postoperatively)
  Each PaO₂ measurement will be reported separately.
Arterial Partial Pressure of Carbon Dioxide (PaCO₂) at Selected Perioperative Time Points (mmHg) | From 10 minutes before anesthesia induction to 45 minutes postoperatively
  Arterial blood gas samples will be collected at the following perioperative time points to measure partial pressure of carbon dioxide (PaCO₂):
  T0 (before anesthesia induction) T1 (10 minutes after induction) T2 (2 minutes after Trendelenburg positioning) T3 (2 minutes after carbon dioxide (CO₂) insufflation) T4 (1 hour after CO₂ insufflation) T5 (2 hours after CO₂ insufflation) T6 (3 hours after CO₂ insufflation) T7 (2 minutes after CO₂ desufflation) T8 (2 minutes after return to supine position) T9 (45 minutes postoperatively)
  Each PaCO₂ measurement will be reported separately.
Arterial Blood pH at Selected Perioperative Time Points | From 10 minutes before anesthesia induction to 45 minutes postoperatively.
  Arterial blood gas samples will be collected at the following perioperative time points to measure blood pH:
  T0 (before anesthesia induction) T1 (10 minutes after induction) T2 (2 minutes after Trendelenburg positioning) T3 (2 minutes after carbon dioxide (CO₂) insufflation) T4 (1 hour after CO₂ insufflation) T5 (2 hours after CO₂ insufflation) T6 (3 hours after CO₂ insufflation) T7 (2 minutes after CO₂ desufflation) T8 (2 minutes after return to supine position) T9 (45 minutes postoperatively) Each pH measurement will be reported separately.
Arterial Bicarbonate (HCO₃-) Level at Selected Perioperative Time Points (mEq/L) | From 10 minutes before anesthesia induction to 45 minutes postoperatively.
  Arterial blood gas samples will be collected at the following perioperative time points to measure bicarbonate (HCO₃-) levels:
  T0 (before anesthesia induction) T1 (10 minutes after induction) T2 (2 minutes after Trendelenburg positioning) T3 (2 minutes after carbon dioxide (CO₂) insufflation) T4 (1 hour after CO₂ insufflation) T5 (2 hours after CO₂ insufflation) T6 (3 hours after CO₂ insufflation) T7 (2 minutes after CO₂ desufflation) T8 (2 minutes after return to supine position) T9 (45 minutes postoperatively)
  Each HCO₃- measurement will be reported separately.
Peak Airway Pressure During Surgery (cmH₂O) | From T1 (10 minutes after anesthesia induction) to T8 (2 minutes after return to supine position).
  Peak airway pressure will be monitored intraoperatively using the Mindray WATO EX-65 anesthesia machine. Measurements will be recorded throughout the surgical procedure (from anesthesia induction to end of anesthesia).
  T1 (10 minutes after induction) T2 (2 minutes after Trendelenburg positioning) T3 (2 minutes after carbon dioxide (CO₂) insufflation) T4 (1 hour after CO₂ insufflation) T5 (2 hours after CO₂ insufflation) T6 (3 hours after CO₂ insufflation) T7 (2 minutes after CO₂ desufflation) T8 (2 minutes after return to supine position)
  Each measurement will be reported separately.
Positive End-Expiratory Pressure (PEEP) During Surgery (cmH₂O) | From T1 (10 minutes after anesthesia induction) to T8 (2 minutes after return to supine position).
  Positive end-expiratory pressure (PEEP) will be monitored intraoperatively using the Mindray WATO EX-65 anesthesia machine. Measurements will be recorded throughout the surgical procedure (from anesthesia induction to end of anesthesia).
  T1 (10 minutes after induction) T2 (2 minutes after Trendelenburg positioning) T3 (2 minutes after carbon dioxide (CO₂) insufflation) T4 (1 hour after CO₂ insufflation) T5 (2 hours after CO₂ insufflation) T6 (3 hours after CO₂ insufflation) T7 (2 minutes after CO₂ desufflation) T8 (2 minutes after return to supine position)
  Each measurement will be reported separately.
Plateau Pressure During Surgery (cmH₂O) | From T1 (10 minutes after anesthesia induction) to T8 (2 minutes after return to supine position).
  Plateau pressure will be monitored intraoperatively using the Mindray WATO EX-65 anesthesia machine. Measurements will be recorded throughout the surgical procedure (from anesthesia induction to end of anesthesia).
  T1 (10 minutes after induction) T2 (2 minutes after Trendelenburg positioning) T3 (2 minutes after carbon dioxide (CO₂) insufflation) T4 (1 hour after CO₂ insufflation) T5 (2 hours after CO₂ insufflation) T6 (3 hours after CO₂ insufflation) T7 (2 minutes after CO₂ desufflation) T8 (2 minutes after return to supine position)
  Each measurement will be reported separately.
Dynamic Pulmonary Compliance During Surgery (mL/cmH₂O) | From T1 (10 minutes after anesthesia induction) to T8 (2 minutes after return to supine position).
  Dynamic pulmonary compliance will be monitored intraoperatively using the Mindray WATO EX-65 anesthesia machine. Measurements will be recorded throughout the surgical procedure.
  T1 (10 minutes after induction) T2 (2 minutes after Trendelenburg positioning) T3 (2 minutes after carbon dioxide (CO₂) insufflation) T4 (1 hour after CO₂ insufflation) T5 (2 hours after CO₂ insufflation) T6 (3 hours after CO₂ insufflation) T7 (2 minutes after CO₂ desufflation) T8 (2 minutes after return to supine position)
  Each measurement will be reported separately.

IPD SHARING:
Plan to Share IPD: No